CLINICAL TRIAL: NCT03001921
Title: Wise Practice of Chinese Hemodialysis (WISHES)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: WISHES
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Haemolyses and Related Conditions
Keywords: Hemodialysis; Patient survival; Quality of life; Hemodialysis access
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — he serum, urine, and DNA will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients: End stage renal disease patients receiving hemodialysis treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Registration of all HD patients in the First Affiliated Hospital of Sun Yat-sen University and other hospital which have signed the contract in China.

SUMMARY:
The investigators are registering all HD patients at recruited hospitals and developing a HD database in China. Patients will be follow-up every 3 months, and both baseline and follow-up information will be entered into the registration system. The patient survival, technical survival, patency rate of access, quality of life and residual renal function for HD patients will be compared using the HD database.

DETAILED DESCRIPTION:
The investigators are registering all end stage renal disease (ESRD) patients receiving hemodialysis (HD) treatment, and developing a HD database in China. Patients' demographic characteristics (including age, gender, height, weight, BMI, smoking, drinking, and education), clinical characteristics (including systolic blood pressure, diastolic blood pressure, primary cause of ESRD, and lab measurements of serum, urine, and access patency), complications, drug information and scores of quality of life at the baseline will be collected. Patients will be follow-up every 3 month, the demographic and clinical characteristics, complications and drug information of patients will be collected at each visit. The investigators also record the outcome at each visit, such as mortality (including all-cause mortality and cardiovascular disease mortality), technical survival, kidney transplantation, transfer to peritoneal dialysis, hospitalization, access failure，etc. The patient survival, technical survival, patency rate of access, quality of life and residual renal function for HD patients will be compared using the HD database.

ELIGIBILITY:
Inclusion Criteria:

End stage renal disease patients receiving hemodialysis treatment.

Exclusion Criteria:

No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage renal disease patients receiving hemodialysis treatment
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2013-12; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient survival of HD patients | 10 years

SECONDARY OUTCOMES:
Quality of life evaluated using SF36 scale for HD patients | 10 years
Patency rate of access for HD patients | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes